CLINICAL TRIAL: NCT04267549
Title: Efficacy and Safety of Conversion Therapy With Sintilimab in Combination With Chemotherapy and Apatinib in Patients With Stage IV Gastric Cancer
Brief Title: Conversion Therapy of Sintilimab in Combination With Apatinib and Chemotherapy in Stage IV Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E20207
Record Dates: First submitted 2020-01-21; First posted 2020-02-13 (Actual); Last update posted 2023-07-06 (Actual); Status verified 2023-05

CONDITIONS: Gastric Cancer Stage IV
Keywords: PD-1 inhibitor; conversion therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — sintilimab; apatinib; S 1 (combination); Taxes

STUDY DESIGN:
Intervention Model Description: eligible patients will be given treatment of sintilimab, apatinib and chemotherapy (nab-paclitaxel) every 3 weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- treatment (Experimental): Eligible patients will be given sintilimab(200mg iv, day 1), apatinib(250mg,once daily), S-1 (60mg, twice daily, day1-14) and nab-paclitaxel(without peritoneal metastases: 260 mg/m^2 iv for 3h; with peritoneal metastases: 200mg/m^2 iv plus 60mg/m^2 ip; day 1) every 3 weeks for at least 3 cycles.
  The feasibility of surgery will be evaluated by a multidisciplinary team every 2-4 cycles.
  Patients assessed as inoperable will be allowed to continue maintenance therapy with the original regimen until disease progression or intolerable toxicity. For patients assessed as operable, apatinib will be discontinued and one more cycle of sintilimab combined with S-1 and nab-paclitaxel will be administered; radical surgery will be performed within 2-4 weeks after the end of treatment.
  Safety run-in stage will be set in the first 6 patients to determine the safety. The study will be terminated if dose-limiting toxicities (DLTs) occur in more than 2 patients.
  Interventions: Drug: sintilimab; Drug: apatinib; Drug: S1; Drug: Nab paclitaxel

INTERVENTIONS:
Drug: sintilimab — a checkpoint inhibitor via blocking PD-1 (programmed cell death-1) site of signaling.
  Other Names: Tyvyt
Drug: apatinib — a multi-target anti-angiogenic tyrosine kinase inhibitor (TKI)
Drug: S1 — S-1 is an oral fluoropyrimidine consisting of tegafur (a prodrug that is converted to fluorouracil, mainly in liver microsomes but also in tumour tissue), gimeracil (an inhibitor of dihydropyrimidine dehydrogenase, which degrades 5-FU), and oteracil (which inhibits the phosphorylation of 5-FU in the gastrointestinal tract, thereby reducing the toxic effects of 5-FU in the intestinum).
Drug: Nab paclitaxel — Nab paclitaxel is a albumin-bound well tolerated paclitaxel than traditional paclitaxel

SUMMARY:
This is a single-arm, phase II study aiming to evaluate the feasibility and efficacy of sintilimab (PD-1 inhibitor) in combination of apatinib and two-drug chemotherapy (S-1 plus nab-paclitaxel) as conversion therapy in patients with stage IV gastric cancer in China.

ELIGIBILITY:
Inclusion Criteria:

* gastric adenocarcinoma confirmed by gastroscopy and pathology (histologically/cytologically ) ;
* life expectancy of ≥3-month；
* unresectable patients who were initially diagnosed as stage IV (clinical stage, American Joint Committee on Cancer 8th edition);
* Eastern Cooperative Oncology Group performance status: 0-1;
* must have at least 1 of the following unresectable factors indicated by CT, MRI or positron emission tomography(PET)-CT:

  1. N3 lymphatic metastasis;
  2. Extensive or bulky lymph nodes;
  3. T4b;
  4. Hepatic metastasis: ≤5 lesions, total diameter of ≤8cm;
  5. Peritoneal metastasis (CY1, P1);
  6. Kukernburg tumor;
* adequate organ function;
* pregnant test negative of females of childbearing potential , and willing to use adequate contraception;
* written Informed Consensus Form;

Exclusion Criteria:

* prior use of any checkpoint inhibitor treatment, including PD-1, programmed cell death ligand-1(PDL-1), CTLA4 etc;
* Her-2 positive with willing to use herceptin treatment;
* prior active autoimmune disease or history of autoimmune disease;
* clinically significant cardiovascular and cerebrovascular diseases, including but not limited to severe acute myocardial infarction within 6 months before enrollment, unstable or severe angina, or coronary artery bypass surgery, Congestive heart failure (New York heart association (NYHA) class > 2), ventricular arrhythmia which need medical intervention, left ventricular ejection fraction(LVEF) < 50%;
* not controlled hypertension;
* prior systemic treatment to metastatic disease；
* previous digestive tract bleeding history within 3 months or evident gastrointestinal bleeding tendency;
* history of immunodeficiency including seropositivity for human immunodeficiency virus (HIV), or other acquired or congenital immune-deficient disease, or active hepatitis ;
* patients who may receive vaccination during study period;
* mental disorders history, or psychotropic drug abuse history;
* unable to orally administration;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-08-30 (Estimated)

PRIMARY OUTCOMES:
R0-surgery conversion rate | up to one year
  The proportion of participants who underwent R0 surgery among all participants.

SECONDARY OUTCOMES:
objective response rate (ORR) | up to one year
  The proportion of participants who achieved complete response(CR) or partial response(PR) per Response Evaluation Criteria in Solid Tumors criteria (RECIST v1.1).
disease control rate (DCR) | up to one year
  The proportion of participants who achieved CR, PR or stable disease(SD) per RECIST v1.1.
conversion rate | up to one year
  The proportion of participants who underwent surgery among all participants.
overall survival (OS) | up to two years
  The time from the first dose of the study treatment to death from any cause.
event-free survival (EFS) | up to two years
  The time from the first dose of the study treatment to any of the following events: progression of disease, local or distant recurrence, or death due to any cause.
Treatment-Related Adverse Events (TRAEs) | from the first day of treatment until 1 month after the end of treatment
  The grade and proportion of participants who experienced TRAEs per National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03
surgery-related complications | from the day of surgery to 30 days postoperatively
  Incidence and grade of surgery-related complications as assessed byper the Clavien-Dindo classification

OTHER OUTCOMES:
pathological response | up to one year after surgery
  Pathological response of the primary tumor was graded according to tumor regression grade (TRG) as follows: 0. (CR), no viable cancer cells, including lymph nodes; 1. (near CR), single cells or rare small groups of cancer cells; 2. (PR), residual cancer cells with evident tumor regression but more than single cells or rare small groups of cancer cells; and 3. (poor or no response), extensive residual cancer with no evident tumor regression.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Gastric Surgery, Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China